CLINICAL TRIAL: NCT02602847
Title: Study of cccDNA in Liver Transplant Patients With B Virus Markers
Brief Title: Study of Covalently Closed Circular DNA (cccDNA) in Liver Transplant Patients With B Virus Markers
Acronym: ECOGREFFE-B
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2012.720
Record Dates: First submitted 2015-11-05; First posted 2015-11-11 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Liver Transplantation
Keywords: Liver transplantation; HBV; cccDNA

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with alcoholic or hepatitis C virus related disease: cccDNA assay on liver biopsy in patients with liver transplantation for alcoholic disease or hepatitis C virus (HCV) related disease, without contact with HBV
  Interventions: Biological: cccDNA assay on liver biopsy
- Hepatitis B core antibody positive donors: cccDNA assay on liver biopsy in patients who receive liver from hepatitis B core antibody positive donors
  Interventions: Biological: cccDNA assay on liver biopsy
- HBV patients: cccDNA assay on liver biopsy in patient with liver transplantation for chronic hepatitis B, with or without HBV replication
  Interventions: Biological: cccDNA assay on liver biopsy

INTERVENTIONS:
Biological: cccDNA assay on liver biopsy — cccDNA assay will be performed on liver biopsies at different times : During transplantation : Liver biopsy of explant and graft and virological biology Between M1 to M3 after transplantation : Liver biopsy between 1 to 3 months after transplantation M12 : Liver biopsy 12 months after transplantation

SUMMARY:
The aim of this study is to validate in the context of liver transplantation, the interest of the cccDNA assay technique developed by the team of Professor Zoulim (INSERM U1052) on liver biopsy and correlate this assay cccDNA in hepatitis B virus (HBV) viral load and serum liver through several groups of patients at transplantation (on graft and native liver explant) and after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patient registered on the national Organ Transplant Waiting List for liver transplantation
* Indication of transplantation :
* Alcoholic related disease without serum anti-hepatitis B core antibody (HBc) (less than 4 weeks) OR - HCV related disease without serum anti-HBc antibody (less than 4 weeks) OR - Patients who sign consent for liver transplantation from hepatitis B core antibody positive donors OR - HBV related disease with positive serum HBs antigen (with or without HBV replication measured by polymerase chain reaction (PCR) within 6 months prior transplantation)
* Signed consent form
* Patient with a social cover
* Patient not covered by any measure of legal protection

Exclusion Criteria:

* Co-infection with HIV, hepatitis delta virus (HDV), HBV (for control arm), HCV (for Test arm) - Positive serology within the4 weeks before inclusion
* Patient covered by any measure of legal protection
* informed consent not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver transplantation planned
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
cccDNA rate on native explant and liver transplant during transplantation and on liver biopsy | 1 year after transplantation
  cccDNA rate will be assessed on native explant and liver transplant during transplantation and on liver biopsy (between M1 to M3 and 12 months (M12) after transplantation) to study the colonization of new hepatocytes by HBV

SECONDARY OUTCOMES:
Correlation between cccDNA rate and serologic status | 1 year after transplantation
  Correlation of cccDNA rate with serologic and virologic status (AgHBe, HBV DNA, ...) at the moment of the transplantation and during post-transplantation period and HBV recurrence
Correlation between cccDNA rate and virologic status | 1 year after transplantation
  Correlation of cccDNA assay with serologic and virologic status (AgHBe, HBV DNA, ...) will be assessed at the moment of the transplantation and during post-transplantation period and HBV recurrence
Correlation between cccDNA rate and patient's treatment | 1 year after transplantation
  Correlation of cccDNA rate with patients' treatments will be assessed at the moment of the transplantation and during post-transplantation period and HBV recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Fabien ZOULIM, MD, PhD, Principal Investigator — Service d'Hépatologie, Hôpital Croix-Rousse, Hospices Civils de Lyon
Locations (5):
- France (5):
  - CHU Grenoble, La Tronche
  - Service d'Hépatologie, Hôpital de la Croix-Rousse, Lyon
  - Hôpital Saint Eloi, Montpellier
  - CHU de Nice, Nice
  - Hôpital Paul Brousse, Villejuif

REFERENCES:
- [Derived] Testoni B, Scholtes C, Plissonnier ML, Paturel A, Berby F, Facchetti F, Villeret F, Degasperi E, Scott B, Hamilton A, Heil M, Lampertico P, Levrero M, Zoulim F. Quantification of circulating HBV RNA expressed from intrahepatic cccDNA in untreated and NUC treated patients with chronic hepatitis B. Gut. 2024 Mar 7;73(4):659-667. doi: 10.1136/gutjnl-2023-330644. PMID 37879886
- [Derived] Villeret F, Lebosse F, Radenne S, Samuel D, Roche B, Mabrut JY, Leroy V, Pageaux GP, Anty R, Thevenon S, Ahmed SS, Hamilton A, Heil M, Scholtes C, Levrero M, Testoni B, Zoulim F; ECOGREFFE Study Group. Early intrahepatic recurrence of HBV infection in liver transplant recipients despite antiviral prophylaxis. JHEP Rep. 2023 Mar 10;5(6):100728. doi: 10.1016/j.jhepr.2023.100728. eCollection 2023 Jun. PMID 37122357